CLINICAL TRIAL: NCT03117712
Title: Influence of Cerebral Blood Supply During Cardiopulmonary Bypass on the Incidence of Postoperative Delirium in Open-heart Surgery
Brief Title: Cerebral Blood Supply During Cardiopulmonary Bypass
Status: Completed | Type: Observational
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Ulrike Weber, Ass.Prof.Dr., Medical University of Vienna
Other Study IDs: 1964/2016
Record Dates: First submitted 2017-04-06; First posted 2017-04-18 (Actual); Last update posted 2019-03-06 (Actual); Status verified 2019-03

CONDITIONS: Postoperative Delirium
Keywords: cerebral blood supply; cardiopulmonary bypass; open-heart cardiac surgery
MeSH Terms: conditions — Emergence Delirium | interventions — Ultrasonography, Doppler, Transcranial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Delirium: patients who develop postoperative delirium after surgery with cardiopulmonary bypass measured by Delirium scores (CAM-ICU, ICDSC), TCD for detection of HITS and carotis duplex sonography
  Interventions: Diagnostic Test: Delirium Scores; Diagnostic Test: Carotis duplex sonography; Diagnostic Test: TCD for detection of HITS
- No delirium: patients who develop no postoperative delirium after surgery with cardiopulmonary bypass measured by delirium scores (CAM-ICU, ICDSC), TCD for detection of HITS and carotis duplex sonography
  Interventions: Diagnostic Test: Delirium Scores; Diagnostic Test: Carotis duplex sonography; Diagnostic Test: TCD for detection of HITS

INTERVENTIONS:
Diagnostic Test: Delirium Scores — * Confusion Assessment method for the ICU (CAM-ICU) and
  * The Intensive Care Delirium Screening Checklist (ICDSC)
  Delirium Scores will be measured at the following timepoints:
  1. Postoperative day (POD) 1
  2. POD 2
  3. POD 5
Diagnostic Test: Carotis duplex sonography — Carotis duplex sonography for perfusion flow will be evaluated at the following timepoints:
  1. Before induction of anaesthesia
  2. Before going on cardiopulmonary bypass (CBP)
  3. During CPB, 5 min after aortic cross clamping
  4. After CPB
  5. 24 hours after CPB
Diagnostic Test: TCD for detection of HITS — Transcranial Doppler ultrasound (TCD) for detection and differentiation of high-intensity transient signals (HITS) in both middle cerebral arteries (MCAs) into artefacts, solid, and gaseous cerebral microemboli (CME) will be performed at the following timepoints:
  1. During cannulation of the ascending aorta
  2. After aortic cross-clamp
  3. After opening of the aortic cross-clamp
  4. During decannulation

SUMMARY:
Postoperative delirium is an acute and fluctuating state of confusion and disorientation with an incidence of 25-70% after cardiac surgery. Possible reasons for this multifactorial complication are hypoperfusion, cerebral microembolization and inflammatory response, which eventually lead to regional or global imbalance between cerebral oxygen demand and supply. Adequate cerebral blood supply depends sufficient blood supply via the vertebral arteries and the internal carotid arteries. The aim of this preliminary study is to investigate if patients who develop delirium after open-heart surgery show differences in their cerebral blood flow during cardiopulmonary bypass (CPB) in extracerebral arterial vessels compared to those patients without delirium.

DETAILED DESCRIPTION:
Postoperative delirium is an acute and fluctuating state of confusion and disorientation, characterized by changes in attention, cognition, consciousness, and perception, with an incidence of 25-70% after cardiac surgery. Possible reasons for this multifactorial complication are hypoperfusion, cerebral microembolization and inflammatory response, which eventually lead to regional or global imbalance between cerebral oxygen demand and supply. This frequent cerebral injury has detrimental and long-lasting consequences and remains a serious healthcare burden, particularly due to its association with higher medical costs, increased morbidity, long-term cognitive deficits, and greater mortality. Progress in reducing the incidence of delirium has been hindered by the lack of a full understanding of its pathophysiology.

Adequate cerebral blood supply depends sufficient blood supply via the vertebral arteries and the internal carotid arteries. Whereby the blood supply of the brain by the carotid arteries is two-thirds and is easily accessable for blood flow examination with Doppler ultrasound.

The aim of this preliminary study is to investigate if patients who develop delirium after open-heart surgery show differences in their cerebral blood flow during cardiopulmonary bypass (CPB) in extracerebral arterial vessels compared to those patients without delirium. Additionally we want to investigate the influence of cerebral microembolisation and CPB associated inflammation in those patients. As secondary outcome measure we also want to determine differences in length of stay (LOS) in the intensive care unit (ICU) as well as in hospital LOS and 30-day mortality.

Methods:

Design:

Prospective observational study

Population:

Elective cardiac surgical patients undergoing valve replacement/reconstruction surgery on cardiopulmonary bypass.

Procedure:

Patients will be enrolled the day before surgery by one physician of the study group.

Anaesthesia will be induced with propofol (1.0-1.5 mg/kg), fentanyl (3-10 μg/kg), and cisatracurium (0.2 mg/kg). It will be maintained with sevoflurane (target BIS value 40-50) 11, and fentanyl (0.05-0.1 μg/kg/min). Patients will receive tranexamic acid (10 mg/kg after anaesthesia induction plus the same dosage in the CPB prime), depending on their kidney function.

Anticoagulation will be achieved with heparin (400 IE/kg) to an activated clotting time (ACT) >400 s.

CPB will be performed using non-pulsatile target flow of 100% calculated cardiac output. Mean arterial pressure will be maintained between 60 to 70 mmHg throughout CPB.

To standardize the intraoperative course of our patients we will limit the intraoperative haematocrit to 22% and the PaCO2-concentration between 30 and 40 mmHg.12 Blood glucose levels will be held between 80-150 mg/dl intra- and postoperatively. Sedation on ICU will be performed using propofol until extubation

Carotis duplex sonography for perfusion flow will be evaluated at the following timepoints:

1. Before induction of anaesthesia
2. Before going on CBP
3. During CPB, 5 min after aortic cross clamping
4. After CPB
5. 24 hours after CPB Blood flow will be derived from the product of the vessels' cross-sectional area and the intensity-weighted mean blood flow velocity through the vessel using a pulsed-wave Doppler in ml/min. Because the sample volume will be adjusted to the width of the vessel at the point where the diameter width will be measured, the measurement can be performed independent of flow conditions (laminary or pulsatile). Imaging of the vessel will be performed in the longitudinal plane, the cross-sectional area will be assumed to be circular.

To diagnose postoperative delirium two delirium assessement tests will be used:

* Confusion Assessment method for the ICU (CAM-ICU) and
* The Intensive Care Delirium Screening Checklist (ICDSC)

Delirium Scores will be measured at the following timepoints:

1. Postoperative day (POD) 1
2. POD 2
3. POD 5

The CAM-ICU will be assessed twice a day (in the morning and in the evening). The Confusion Assessment Method (CAM) will be performed after discharge from the ICU.

Transcranial Doppler ultrasound (TCD) for detection and differentiation of high-intensity transient signals (HITS) in both middle cerebral arteries (MCAs) into artefacts, solid, and gaseous cerebral microemboli (CME) will be performed at the following timepoints:

1. During cannulation of the ascending aorta
2. After aortic cross-clamp
3. During decannulation All collected data will be saved password-protected in an electronic database on the department's server after data collection has been finished. Only studyteam-members will have access to this data. After completion of the study the results are to be published according to GCP-standards.

ELIGIBILITY:
Inclusion Criteria:

elective cardiac surgery valve replacement/reconstruction cardiopulmonary bypass

Exclusion Criteria:

* Emergency procedures
* Postoperative need for extracorporal cardiac assist device
* Untreated or uncontrolled arterial hypertension
* Profound hypothermic CPB (body temperature <34°C)
* History of preoperative dementia
* History of Stroke
* Significant carotid artery stenosis
* Age < 18 years
* Chronic renal replacement therapy
* Declined informed consent

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Elective cardiac surgical patients undergoing valve replacement/reconstruction surgery on cardiopulmonary bypass.
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
cerebral blood flow | during surgery
  Differences in mean laminar cerebral blood flow on cardiopulmonary bypass during open heart surgery between patients with and without postoperative delirium

SECONDARY OUTCOMES:
HITS (high-intensity transient signals) | during surgery
  Difference in the number and quality of HITS measured with transcranial Doppler ultrasound between patients with and without delirium

CONTACTS AND LOCATIONS:
Overall Officials: Ulrike Weber, M.D., Principal Investigator — Medical University of Vienna
Locations (1):
- Medical university of vienna, General hospital of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No